CLINICAL TRIAL: NCT06643611
Title: Addressing Disparities in Diabetes Care: Integrating Continuous Glucose Monitors and Pharmacist Medication Management for Uninsured Racial Minority Patients
Brief Title: Addressing Disparities in Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Society of Health-System Pharmacists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00115753
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Glucose Monitor (Experimental): Patients in the intervention arm will receive a continuous glucose monitor in addition to usual care. These patients will be scheduled at least once monthly for clinical pharmacy visits.
  Interventions: Behavioral: Continuous Glucose Monitor
- Usual Care (Active Comparator): Patients in the usual care arm will have routine physician office visits every 3 months if HbA1c outside goal or every 6 months if HbA1c within goal. Medication regimens will be managed by physicians, nurse practitioners, and physician assistants.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Continuous Glucose Monitor — Patient will be provided a continuous glucose monitor. Pharmacist will provide information regarding how to best manage type 2 diabetes.
  Arms: Continuous Glucose Monitor
Behavioral: Usual Care — Routine physician office visits and hemoglobinA1c every 3 for those with HbA1c outside goal and every 6 months for those with HbA1c within goal. Medication regimens managed by physicians, nurse practitioners, and physician assistants. Patients are sent reminders on the phone prior to their visits or when they are due for a visit or any physical examination.
  Arms: Usual Care

SUMMARY:
The purpose of this research is to find out if using a continuous glucose monitor and working with a clinical pharmacist can help improve the health of uninsured minority patients with type 2 diabetes.

DETAILED DESCRIPTION:
The objective of this research is to determine the effectiveness of a targeted intervention that integrates continuous glucose monitors and pharmacist-led comprehensive medication management services among uninsured adult patients with poor glycemic control on basal insulin, specifically focusing on Black and Hispanic populations. This pilot study is designed to help justify implementing this intervention on a larger scale within our healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic or non-Hispanic Black
* Diagnosis of Type 2 diabetes
* HbA1c ≥8% within the past 3 months
* Active prescription for insulin and injecting at least 1 time daily

Exclusion Criteria:

* Gestational diabetes
* Type 1 diabetes
* Receiving care by endocrinologist
* Continuous glucose monitor use within the past 6 months
* Receiving long term, hospice, or palliative care services
* Malignant cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c | Baseline to Month 6
  Change in percentage for Hemoglobin A1c. Normal range for hemoglobin A1c is 4.2%-14%. A low level indicates no diabetes and a high level indicates uncontrolled diabetes.

SECONDARY OUTCOMES:
Appraisal of Diabetes Scale | Baseline, 1 Month Post Intervention
  Health-related quality of life will be measured using Appraisal of Diabetes scale (ADS). The ADS is a diabetes-specific quality of life instrument. It consists of 7 items on how diabetes affects the respondent. The score of each item ranges from 0 to 5 with 0 representing the least effect of diabetes and 5 the greatest effect of diabetes. The total score is calculated by summing the scores of individual items.
Diabetes Treatment Satisfaction Questionnaire | Baseline, 1 Month Post Intervention
  Treatment satisfaction will be measured using the Diabetes Treatment Satisfaction Questionnaire (DTSQ). The DTSQ includes eight items on satisfaction with diabetes treatment, convenience, flexibility, understanding of diabetes, possibility of continuation of the current treatment and recommendation to others. Each item is scored on a scale from 0 to 6, with higher score indicating higher satisfaction.
Change in Medication Adherence | 6 Months Post Intervention
  Medication adherence will be determined from prescription fill data and reported in the form of medication possession ratio (the sum of days of supply during a time period divided by the number of days in that time period). The change during six months before and after intervention start (time of assessment of study criteria for the control group) will be reported.
Number of Hours Glucose Level in Normal Range | Week 1 and 2 of intervention, Last Two Weeks of Intervention
  Number of hours patient's glucose level is within normal range of 70-100.
Number of Hours Glucose Level Above Normal Range | Week 1 and 2 of intervention, Last Two Weeks of Intervention
  Number of hours patient's glucose level is above normal range of 70-100.
Number of Hours Glucose Level Below Normal Range | Week 1 and 2 of intervention, Last Two Weeks of Intervention
  Number of hours patient's glucose level is below normal range of 70-100.
Average Glucose Level | Week 1 and 2 of intervention, Last Two Weeks of Intervention
  Average glucose level during the first two weeks of intervention. Normal range is 70-100 mg/dL. A low-level average indicates good glycemic control. A high level indicates uncontrolled diabetes.
Glucose Management Indicator Percentage | Week 1 and 2 of intervention, Last Two Weeks of Intervention
  The glucose management indicator is an updated approach for estimating hemoglobin A1c from continuous glucose monitoring data. Range is 5.7%-14%.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Larson, PharmD, CPP, Principal Investigator — Myers Park Internal Medicine
Locations (1):
- Atrium Health Myers Park Internal Medicine Clinic, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT06643611/ICF_000.pdf